CLINICAL TRIAL: NCT07291128
Title: Effects of VOJTA Technique on Muscle Tone, Gross Motor Function and Balance on Ataxic Cerebral Palsy.
Brief Title: Effects of VOJTA Technique on Ataxic Cerebral Palsy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/043 Fareeha
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ataxic Cerebral Palsy
Keywords: vojta; muscle tone; ataxic cerebral palsy; gross motor function; balance
MeSH Terms: conditions — Cerebral Palsy, Ataxic, Autosomal Recessive

STUDY DESIGN:
Intervention Model Description: After recruitment of participants into study they will be allocated to their respective groups utilizing the online randomizer tool.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1/ VOJTA (Experimental): Participants in this arm will receive VOJTA reflex locomotion therapy, which involves activating innate locomotor patterns through manual stimulation of specific pressure zones while the child is positioned in standardized postures. This arm examines the effectiveness of VOJTA therapy in improving muscle tone, balance, and gross motor function in children with ataxic cerebral palsy
  Interventions: Behavioral: VOJTA
- Group 2 / Conventional Physical Therapy (Active Comparator): Participants in this arm will receive routine conventional physiotherapy commonly used for cerebral palsy rehabilitation. This includes Neurodevelopmental Therapy (NDT/Bobath-based methods), balance training, core strengthening, stretching, and functional task-oriented exercises. This arm serves as the comparison group.
  Interventions: Behavioral: Conventional Physical Therapy

INTERVENTIONS:
Behavioral: VOJTA — VOJTA therapy will be administered by a physiotherapist. The intervention involves mechanical stimulation of defined reflex zones located on the trunk and limbs while the child is in prone, supine, or side-lying postures. Stimulation elicits automatic reflex creeping or reflex rolling patterns that enhance trunk activation, postural control, coordination, and normalization of muscle tone. Treatment follows the standardized VOJTA protocol, applying precise direction, pressure, and duration of stimulation. The frequency will be 5 sessions per week for 8 weeks with duration of 30 minutes.
  Arms: Group 1/ VOJTA
Behavioral: Conventional Physical Therapy — Conventional physiotherapy includes evidence-based approaches commonly applied for cerebral palsy rehabilitation. This may include NDT/Bobath principles, balance and postural stability exercises, core strengthening, stretching, functional mobility training, and sensory-motor facilitation. No VOJTA stimulation will be used. All participants follow a standardized treatment protocol to ensure consistency. The frequency will be 5 sessions per week for 8 weeks with duration of 30 minutes.
  Arms: Group 2 / Conventional Physical Therapy

SUMMARY:
Ataxic cerebral palsy (CP) is the least common subtype of CP and it is primarily caused by cerebellar damage that results in hypotonia, impaired balance, poor coordination, tremors, wide-based gait, and significant difficulties in trunk stability and uncontrolled movements. These impairments greatly affect functional mobility and independence in life. This randomized controlled trial aims to evaluate the effects of VOJTA therapy on muscle tone, gross motor function, and postural control in children with ataxic CP aged 2-6 years. VOJTA therapy is based on reflex locomotion, which activates innate central motor programs by stimulating specific pressure zones in defined positions, potentially improving postural alignment and coordinated muscle activation. A total of 40 children will be randomly assigned to either the VOJTA therapy group or a conventional physiotherapy group. Both groups will receive total of 5 sessions per week for 8 weeks and the Outcomes will be measured at baseline, 4 weeks, and 8 weeks using the Modified Ashworth Scale (MAS) for muscle tone, Gross Motor Function Measure (GMFM-88) for gross motor function and Pediatric balance scale for for balance. This study hypothesizes that VOJTA therapy will produce greater improvements in muscle tone, gross motor function and balance as compared to conventional physical therapy techniques. Findings may support evidence-based rehabilitation strategies for ataxic CP and contribute to improved functional independence and quality of life in this understudied population.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a lifetime neurological condition caused by an early injury to the brain that cannot change over time, and although the brain injury itself is non-progressive, the motor problems can be different as they grow CP really affects the whole body movement, and the things that are performed by the body's muscles like, posture, coordination, muscle tone, and balance, In other cases, however, sensory processing challenges are present along with these and the child may experience delayed motor development. Among the different types of CP, ataxic cerebral palsy is the one that occurs least often, with an incidence of only around 5-10% of total CP cases. Although it is a type of cerebral palsy that is complex and therefore, more debilitating. The defining feature of ataxic CP which is mainly due to the cerebellar part of the brain being affected and motor commands of the body being uncoordinated and imprecise. Children affected by this type of CP usually have hypotonia, tremors when trying to perform a task, dysmetria, are unsteady or walk with feet far apart, have poor control of the upper body and reach motor skills later than the typical child, therefore every movement that they try to make, including the most basic ones like sitting, reaching, standing or walking, are very hard. Especially, the very important motor and communication functions of the hands, arms, and legs are affected. But although all of these problems point to a very serious form of CP, ataxic CP has so far gotten far less research attention than spastic CP and consequently, less clinical evidence-based guidance that is tailored specifically to this subtype. Most of the time, children that suffer from ataxic CP are subjected to traditional physiotherapy methods such as Neurodevelopmental Therapy, Bobath techniques, balance training, sensory integration, or strengthening exercises; however, these methods are only moderately successful as they do not directly address the specific coordination and postural control difficulties that are related to cerebellar dysfunction, thus, they do not offer any substantial change in the quality of life of the affected children. Since then the gap has become wider and that is why there is more and more interest in the neurophysiological methods that stimulate and activate the central motor pathways that are responsible for posture and movement. VOJTA therapy, which is also known as reflex locomotion therapy, provides a different method by the activation of movements that are automatic and innate through the specific stimulation of pressure that is applied while the child is in the defined postures. The treatment is thought to activate both spinal and supraspinal pathways thus increasing the muscle activation in the trunk, improving postural control, and causing the brain to generate new pathways. Studies on children suffering from cerebral palsy with spastic condition have reported better results in the areas of gross motor function, trunk stability, and early motor development. Neuroimaging has shown the activation of sensorimotor cortical areas during the stimulation of VOJTA. However, there is not enough research on the VOJTA therapy application for children with ataxic CP although they experience severe coordination and balance problems. This research intends to support filling this important gap by analyzing the VOJTA therapy effect on muscle tonicity, gross motor function, and balance in children aged 2-6 years with ataxic CP. Out of forty participants, some will be placed in the VOJTA therapy group while others will be put in the conventional physiotherapy group and the treatment will be done five times per week for eight weeks. The evaluation of the outcomes will be done at the beginning, after four weeks, and after eight weeks through the Modified Ashworth Scale for muscle tone, the Gross Motor Function Measure for motor performance, and the Pediatric Balance Scale for balance. The hypothesis of the study is that VOJTA therapy will bring about a more significant reduction of the problem in muscle tone, balance, and gross motor functions than conventional physiotherapy. This study, by concentrating on one of the least studied types of CP, has the capacity to help reshape clinical practice, enhance rehabilitation techniques better, and lead to less standard and more evidence-based care for the child with CP.

ELIGIBILITY:
Inclusion Criteria:

Both male and female participants would be included

Children diagnosed with ataxic cerebral palsy.

Age range of participants will be 2 to 6 years old.

Participants included will be at level 2 on gross motor function classification scale.

Participants included will have ATNR reflex.

Stable medical condition for the past three months with no hospitalizations.

Exclusion Criteria:

Presence of severe comorbidities i.e. neurological or orthopedic conditions.

Patients having significant cognitive deficits

Down syndrome, hydrocephalus, epilepsy, autism and medically ill children

Children with visual or auditory deficits affecting postural control and balance assessment.

Ongoing pharmacological treatment (e.g., muscle relaxants or antiepileptic) likely to influence muscle tone or motor function during the study period

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline, 4 weeks, 8 weeks
  Muscle tone will be evaluated using the Modified Ashworth Scale, which measures resistance during passive movement to assess tone abnormalities. Scores range from 0 to 4, with higher scores indicating increased resistance or greater tone abnormality. Improvement is defined as a reduction in MAS scores or normalization of tone patterns following the intervention period.
Gross Motor Function Measure-88 (GMFM-88) | Baseline, 4 weeks, 8 weeks
  Gross motor function will be assessed using the GMFM-88, a validated observational measure designed to evaluate changes in motor skills across five domains (lying/rolling; sitting; crawling/kneeling; standing; walking/running/jumping). Total and domain-specific scores will be analyzed. Improvement is defined as an increase in GMFM-88 scores after the intervention.
Pediatric Balance Scale (PBS) | Baseline, 4 weeks, 8 weeks
  Balance performance will be measured using the Pediatric Balance Scale, which includes 14 tasks assessing static and dynamic balance in functional positions. Scores range from 0 to 56, with higher scores representing better balance control. Improvement is defined as an increase in PBS scores following treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ha SY, Sung YH. Effects of Vojta approach on diaphragm movement in children with spastic cerebral palsy. J Exerc Rehabil. 2018 Dec 27;14(6):1005-1009. doi: 10.12965/jer.1836498.249. eCollection 2018 Dec. PMID 30656162
- [Result] Sanchez-Gonzalez JL, Sanz-Esteban I, Menendez-Pardinas M, Navarro-Lopez V, Sanz-Mengibar JM. Critical review of the evidence for Vojta Therapy: a systematic review and meta-analysis. Front Neurol. 2024 Apr 22;15:1391448. doi: 10.3389/fneur.2024.1391448. eCollection 2024. PMID 38711552